CLINICAL TRIAL: NCT06195657
Title: Pre-video Assisted Thoracoscopy Surgery (VATS) Localization of Ground Glass Solitary Pulmonary Nodules: the Sliding Wire Technique
Brief Title: Pre-operative Localization of Ground Glass Solitary Pulmonary Nodules
Acronym: SLIDINGWIRE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 23Imagerie04
Record Dates: First submitted 2023-12-05; First posted 2024-01-08 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-12

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objectives: The main drawback of the hook-wire technique for locating ground glass nodules before video assisted thoracoscopic surgery (VATS) resection is the risk of the hook dislodging during single lung ventilation as the lung collapses. In order to reduce the friction of the thread in the wall, the investigators modified the technique by first positioning a catheter in the chest wall and introducing the carrying needle through the catheter. The objective was to evaluate the success rate and complications of this technique.

Material and Methods : the investigators retrospectively included all patients undergoing VATS resection of solitary lung nodules after localization using the sliding wire technique.

ELIGIBILITY:
Inclusion Criteria

- All patients who underwent VATS for pulmonary nodule resection in the thoracic surgery department of Nice University hospital after pre-operative hook-wire insertion using the sliding-wire technique

Exclusion criteria: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the university hospital of Nice, France
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2021-11 (Actual); Study Completion 2021-11 (Actual)

PRIMARY OUTCOMES:
Success rate of the procedure | Up to 4 hours
  Percentage of hook wires remaining anchored during the surgical resection of suspect nodules

SECONDARY OUTCOMES:
Complications | Up to 4 hours
  Rate of complication of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Padovani, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU NICE, Nice, Alpes Maritimes, France

IPD SHARING:
Plan to Share IPD: Undecided